CLINICAL TRIAL: NCT06984757
Title: Mid-frontal Delta/Theta and Cognitive Control
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nandakumar Narayanan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Nandakumar Narayanan, Professor of Neurology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 201707828; 2R01NS100849-06A1 (NIH)
Record Dates: First submitted 2025-04-16; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Parkinson&Amp;Amp;#39;s Disease (PD)
Keywords: Parkinson's disease; deep-brain stimulation; mild cognitive impairment; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Deep Brain Stimulation; Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Deep-brain Stimulation (DBS) (Experimental)
  Interventions: Device: Deep-brain Stimulation
- Transcranial Magnetic Stimulation (TMS) (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- Transcranial Alternating Current Stimulation (tACS) (Experimental)
  Interventions: Device: Transcranial Alternating Current Stimulation
- Observational (No Intervention)

INTERVENTIONS:
Device: Deep-brain Stimulation — a neurosurgical procedure that uses implanted electrodes and electrical stimulation to treat movement disorders and certain neuropsychiatric conditions when medications are ineffective or cause significant side effects.
  Arms: Deep-brain Stimulation (DBS)
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a non-invasive treatment that uses magnetic fields to stimulate specific areas of the brain.
  Arms: Transcranial Magnetic Stimulation (TMS)
Device: Transcranial Alternating Current Stimulation — Transcranial Alternating Current Stimulation (tACS) is a non-invasive brain stimulation technique that uses weak, alternating electrical currents applied to the scalp to modulate brain activity and potentially influence cognitive processes by entraining brain oscillations.
  Arms: Transcranial Alternating Current Stimulation (tACS)

SUMMARY:
Abstract Cognitive symptoms of Parkinson's disease (PD) include deficits in attention, working memory, and reasoning. These deficits affect up to 80% of PD patients and lead to mild cognitive impairment (PD-MCI) and dementia in PD (PDD). There is a critical need to better understand cognitive impairment in PD to develop new targeted treatments. The long-term goal is to define the mechanisms of PD-related cognitive impairment. PD involves diverse processes such as dopamine and acetylcholine dysfunction, synuclein aggregation, and genetic factors. During the past funding period, the investigators linked PD-related cognitive impairment to dysfunction in frontal midline delta (1-4 Hz) and theta (5-7 Hz) rhythms, which the work has established as a marker of cognitive control. However, it is unknown why PD patients have deficits in these low-frequency brain rhythms. The preliminary magnetic resonance imaging (MEG) and magnetoencephalography (MRI) implicate the anterior midcingulate cortex (aMCC) as a potential source of frontal midline delta/theta rhythms. In the next funding period, the objective is to determine the mechanisms and predictive power of delta/theta rhythms in PD, which will help to better understand the pathophysiology of PD-related cognitive impairment. Collaboration between the University of New Mexico (UNM) and University of Iowa (UI) that will bring together MEG, MRI, longitudinal EEG, and adaptive subthalamic (STN) deep-brain stimulation (DBS). The investigators will test the overall hypothesis that frontal midline delta/theta dysfunction contributes to cognitive impairments in PD. In Aim 1, the investigators will determine the structural basis for delta/theta rhythm deficits in PD. In Aim 2, the investigators will determine the predictive power of delta/theta rhythm deficits in PD. In Aim 3, the investigators will determine how tuned low-frequency STN DBS impacts cortical activity and cognition. The results will have relevance for basic-science knowledge of the fundamental pathophysiology of cognitive impairment in PD and related dementias. Because this proposal will study patients with PDD, the findings are directly relevant to Alzheimer's-related dementias (ADRD).

DETAILED DESCRIPTION:
Up to 80% of patients with Parkinson's disease (PD) will suffer from cognitive symptoms, including impaired attention, planning, reasoning, and working memory as well as hallucinations, visuospatial dysfunction, and delusions. These impairments lead to mild cognitive impairment (PD-MCI) and dementia (PDD) in PD. Cognitive symptoms of PD are associated with enormous costs to society. There are no clear biomarkers and few effective treatments for PD-MCI/PDD. Because risk for PD increases dramatically with age, this problem will surge as the population grows older. The mechanisms contributing to PD-MCI/PDD are unknown. The investigators have found that low-frequency (1-8 Hz; or delta/theta bands) brain rhythms might be helpful in diagnosing cognitive dysfunction in PD. This delta/theta activity originates from areas of medial frontal cortex, such as the anterior cingulate, and is detectable by mid-frontal scalp EEG electrodes. We have found that mid-frontal delta/theta brain rhythms are engaged when healthy individuals detect novelty, errors, and conflict, or make decisions. These rhythms are attenuated in PD patients. The working model is that PD patients manifest diverse neuronal and network deficits that impair mid-frontal delta/theta activity, leading to failures in engaging cognitive control. These abnormalities contribute to PD-MCI and PDD.

In this proposal, we combine 'big-data' machine learning tools and new brain-stimulation paradigms to investigate the role of mid-frontal delta/theta rhythms in PD. We will test the overall hypothesis that mid-frontal delta/theta impairments are a mechanism of cognitive dysfunction in PD. We will determine if mid-frontal delta/theta activity predicts PD-MCI/PDD and if subthalamic nucleus deep-brain stimulation (DBS) at delta/theta frequencies improves cognitive control in PD patients. Because these experiments involve EEG recordings across several PD patient populations and brain stimulation, each of these aims will provide independent mechanistic insight into cognitive dysfunction in PD. PD is a complex disease, but if cortical EEG abnormalities are a consistent theme, it might inspire new diagnostic tools or new brain-stimulation therapies for cognitive dysfunction in PD. Results from this proposal could also be important for other neurodegenerative diseases such as dementia with Lewy bodies and Alzheimer's disease.

* We will perform the study on Parkinson's disease (PD) patients. PD patient takes anti-Parkinsonian medication (Levodopa) to improve motor symptoms. Medication can change their cognitive performances and neuronal activity; therefore, we will ask (on the phone) patients to withdraw medication (the night before) so that the next morning they will be off medication. For this study, it is crucial that the washout period is >12 hours. During OFF medication, PD patients will only be slow in walking and performing motor activities. There won't be worse effects since it's a motor disorder. We will stop the experiments if the subject worsens during the washout period, and we will provide him/her medications. At the same time, the subject will be examined by the expert neurologist.
* The purpose of the other experiments that are part of this study is to investigate the functions of the specific brain circuit underlying motor and cognitive tasks. Specifically, we are interested in investigating a well-known brain area that allows humans to interrupt ongoing neural representations interacts with active, ongoing motor processes (action initiation and execution) and cognitive processes within the context of simple laboratory tasks. The interaction between neural regions underlying controlling ongoing motor and cognitive processes allows the brain circuit to improve motor action and thought processes when necessary. Typically, patients with Parkinson's disease are slow to execute motor tasks and also show impairment in cognitive performance. We will combine electroencephalography (EEG) with transcranial magnetic stimulation (TMS) to study the effects of stimulation on neuronal activity.

The study will use TMS to temporarily and reversibly alter the activity of a specific node (brain area) of the wider brain network (specifically, the pre-supplementary motor, pre-motor area, and motor cortical regions), and measure the effects of this stimulation-related alteration on neural and behavioral measurements of motor and cognitive tasks. The brain stimulation methods use different protocols of TMS to evoke internally generated neural discharges through the use of focal magnetic fields.

* All subjects will perform questionnaires related to the cognitive and motor impairments.
* Afterwards, we will record EEG and respiratory data during elementary cognitive tasks such as interval timing, oddball detection, stop-signal, and Simon choice reaction-time tasks and upper- and lower limb motor tasks (flexion and extension (such as key board pressing and pedaling), gait imagery, and observation)and at resting state (during sitting (eyes open and close) and standing on soft pad) from PD patients without PD-MCI/PDD, patients with PD-MCI, patients with PDD, and demographically-matched healthy controls. We will also include patients with Alzheimer's disease (AD) and Lewy body dementia (DLB) as control subjects since they don't have dopamine deficiency. We will also include healthy young and middle age adults as comparison groups to compare neural mechanisms of cognitive control across age groups.
* For another aim, we will record EEG with 4 Hz STN DBS during above tasks (rest, cognitive, and motor tasks ) in PD patients.
* For another study, We will record EEG with TMS during simple upper and lower limb flexion-extension motor task (such as key board pressing and pedaling), cognitive tasks (as above) and resting state (as above) in different group of PD subjects. We will not include PD subjects with DBS in TMS experiments. We will recruit PD subjects on different day only for EEG-TMS experiment.
* We will also be piloting the behavioral tasks with a small group of control subjects and PD patients. This will allow us to optimize the tasks to be used in all other aims.
* We would like to use patients with DBS in VIM thalamus for essential tremor as a control.
* For another study, we will record EEG during tasks in healthy young and middle-aged adults. We will be examining brain circuitry and activity involved with cognitive tasks. We will also be acquiring information from the control young adults' mothers about stress experienced while they were pregnant with their child (the control subjects). The purpose of this study is to examine the relationship between prenatal and early life stress and brain function during adulthood.
* For another study, we will record patient quality of life using questionnaires and interviews after EEG recordings have been completed. This information will then be correlated with prior collected EEGs to assess the relationship between EEG and quality of life in PD patients. We will be recruiting approximately 100 parkinson's patients who have already completed EEG recordings and cognitive tasks for the study for the quality of life project. The prior projects indicate that this amount is enough to discern differences in EEG activity in the regions of concern to establish a relationship between this signal and quality of life surveys.
* For another study, we will study the effects of transcranial Alternating Current Stimulation (HD-tACS) on EEG and behavioral responses. We will do EEG recordings in PD patients during cognitive tasks (the flanker task and the N-back task) and resting condition (as above) during and after tACS. We will be recruiting 24 Parkinson's disease patients.

ELIGIBILITY:
We will study individuals with idiopathic mild-moderate Parkinson's Disease. Diagnosis will be confirmed by Dr. Narayanan - a neurologist.

Inclusion criteria:

GROUP 1: Parkinson's disease without cognitive impairment

1. Parkinson's disease, with MOCA > 26
2. under stable PD medication
3. able to walk independently, make their own decisions
4. age range = 18 - 89 years old

GROUP 2: Parkinson's disease with mild cognitive impairment

1. Parkinson's disease, with MOCA 23-26
2. under stable PD medication
3. able to walk independently, make their own decisions
4. age range = 18 - 89 years old

GROUP 3: Parkinson's disease with dementia

1. Parkinson's disease, with MOCA < 23
2. under stable PD medication
3. Make their own decisions
4. age range = 18 - 89 years old

GROUP 4: Parkinson's disease with STN-DBS 1) Parkinson's disease with functioning bilateral STN-DBS electrodes 2) under stable PD medication 3) able to walk independently, make their own decisions 4) age range = 18 - 89 years old 5) THIS GROUP WILL NOT UNDERGO TMS

GROUP 5: Parkinson's disease without DBS and with no seizure history for EEG-TMS study

1. Parkinson's disease with MOCA 23-30
2. under stable PD medication
3. able to walk independently, make their own decisions
4. age range = 18 - 89 years old

GROUP 6: Essential tremor with VIM-DBS

1) Essential tremor with functioning bilateral VIM-DBS electrodes 2) able to walk independently, make their own decisions 3) age range = 18 - 89 years old 4) THIS GROUP WILL NOT UNDERGO TMS

GROUP 7: Parkinson's disease without DBS and with no seizure history for EEG-HD-tACS study 1) Parkinson's disease with MOCA 23-30 2) under stable PD medication 3) able to walk independently, make their own decisions 4) age range = 18 - 89 years old

Exclusion criteria:

Patients with dementia with Lewy Bodies and Alzheimer's disease, drug-induced parkinsonism, Parkinson's-plus, on investigational drugs, with hearing loss will be excluded, or with color-blindness will be excluded. Subjects with a history of neuropsychiatric disorders, like Schizophrenia or Depression will be also be excluded.

For the TMS sub-study, PD patients with DBS leads will be excluded and any subject with a seizure disorder will also be excluded. For the HD-tACS sub-study, PD patients with DBS leads will be excluded and any subject with a seizure disorder will also be excluded.

Control Group: patients with Alzheimer's Disease (AD) and dementia with Lewy Bodies (DLB) A group of patients with AD and DLB will be recruited for the cognitive tasks to compare data with PD. Since AD is non-dopamine deficiency disease so they can serve as another control group for the study.

Inclusion criteria:

1) age range = 18 - 89 years old (will have to match with the age of subjects with Parkinson's Disease)

Exclusion criteria:

1) with any neurological disorders, including epilepsy

Control Group: patients with mTBI A group of patients with mTBI will be recruited for the cognitive tasks to compare data with PD.

Inclusion criteria:

1) age range = 18 - 89 years old (will have to match with the age of subjects with Parkinson's Disease)

Exclusion criteria:

Control Group: patients with 16pDel Autism A group of patients with 16pDel Autism will be recruited for the cognitive tasks to compare data with PD.

Inclusion criteria:

1) age range = 18 - 89 years old (will have to match with the age of subjects with Parkinson's Disease)

Exclusion criteria:

Control Group: patients with Brain Lesions A group of patients with Brain Lesions will be recruited for the cognitive tasks to compare data with PD.

Inclusion criteria:

1) age range = 18 - 89 years old (will have to match with the age of subjects with Parkinson's Disease)

Exclusion criteria:

Control Group: Older Normal Subjects A group of older healthy individuals will be matched with subjects with Parkinson's disease in terms of age, sex, and years of education. We will also recruit a small group of older healthy individuals specifically to pilot new behavioral tasks.

Inclusion criteria:

1) age range = 35 - 99 years old (most of this group will have to match with the age of subjects with Parkinson's Disease. One subset from this group (N = 40) will be independent from the demographics of the subjects with Parkinson's Disease, so they can have a wider age range).

Exclusion criteria:

1) with any neurological disorders, including epilepsy

Control Group: Older Subjects with Mood Disorders A group of older individuals with Mood Disorders will be recruited to perform cognitive tasks to compare data with both PD with Mood Disorders and PD without Mood Disorders.

Inclusion criteria:

1) age range = 18 - 89 years old (will have to match with the age of subjects with Parkinson's Disease)

Exclusion criteria:

1) with any neurological disorders, including epilepsy

Control group: Healthy young and middle-aged adults

* A group of healthy young and middle-aged adults without Parkinson's disease or other neurological issues.
* 1) age range = 18-60 years old
* Exclusion criteria: 1) any neurological disorders, including epilepsy

Control subjects' mothers

- The group of mothers of the healthy young adult control subjects.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 635 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes to EEG physiological parameters (mid-frontal delta/theta activity) due to Parkinson's disease (PD) at Day 1 | From enrollment to the end of treatment at Day 1
  The investigators use a conventional repeated-measures ANOVA where the independent variable is PD/PD-MCI/PDD and the dependent variable is mid-frontal delta/theta activity (EEG physiological parameter).

SECONDARY OUTCOMES:
Changes to EEG physiological parameters (mid-frontal delta/theta activity) due to the Deep Brain Stimulation (DBS) stimulation setting at Day 1 | From enrollment to the end of treatment at Day 1
  The investigators use a conventional repeated-measures ANOVA where the independent variable is the deep brain stimulation (DBS) setting and the dependent variable is mid-frontal delta/theta activity (EEG physiological parameter).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
We may share health information related to this study with other parties including federal government regulatory agencies, the University of Iowa Institutional Review Boards and support staff.
Supporting Information: Study Protocol
Time Frame: 25 Sept 2017 to 31 Dec 2029
Access Criteria: We keep participation in this research study confidential to the extent permitted by law. However, it is possible that other people such as those indicated below may become aware of participation in the study and may inspect and copy records pertaining to this research. Some of these records could contain information that personally identifies the participant.
  * federal government regulatory agencies,
  * auditing departments of the University of Iowa, and
  * the University of Iowa Institutional Review Board (a committee that reviews and approves research studies)
  To help protect confidentiality, we store all information in a locked, password encrypted secure research drive that is stored in a locked room. If we write a report or article about this study or share the study data set with others, we will do so in such a way that you cannot be directly identified.

REFERENCES:
- [Background] Anjum MF, Espinoza AI, Cole RC, Singh A, May P, Uc EY, Dasgupta S, Narayanan NS. Resting-state EEG measures cognitive impairment in Parkinson's disease. NPJ Parkinsons Dis. 2024 Jan 3;10(1):6. doi: 10.1038/s41531-023-00602-0. PMID 38172519
- [Background] Narayanan NS, Jourahmad Z, Cole RC, Cavanagh JF. Cognition falters at ~4 Hz in Parkinson's disease. Trends Cogn Sci. 2024 Sep;28(9):789-791. doi: 10.1016/j.tics.2024.06.002. Epub 2024 Jul 12. PMID 39003229
- [Background] Yeager BE, Twedt HP, Bruss J, Schultz J, Narayanan NS. Salience network and cognitive impairment in Parkinson's disease. medRxiv [Preprint]. 2023 Oct 14:2023.10.13.23296825. doi: 10.1101/2023.10.13.23296825. PMID 37873396
- [Background] Bosch TJ, Cole RC, Bezchlibnyk Y, Flouty O, Singh A. Effects of Very Low- and High-Frequency Subthalamic Stimulation on Motor Cortical Oscillations During Rhythmic Lower-Limb Movements in Parkinson's Disease Patients. J Parkinsons Dis. 2023;13(4):549-561. doi: 10.3233/JPD-225113. PMID 37092236
- [Background] Singh A, Cole RC, Espinoza AI, Wessel JR, Cavanagh JF, Narayanan NS. Evoked mid-frontal activity predicts cognitive dysfunction in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2023 Nov;94(11):945-953. doi: 10.1136/jnnp-2022-330154. Epub 2023 Jun 1. PMID 37263767
- [Background] Lin LC, Cole RC, Greenlee JDW, Narayanan NS. A Pilot Study of Ex Vivo Human Prefrontal RNA Transcriptomics in Parkinson's Disease. Cell Mol Neurobiol. 2023 Aug;43(6):3037-3046. doi: 10.1007/s10571-023-01334-8. Epub 2023 Mar 23. PMID 36952070
- [Background] Anjum MF, Espinoza A, Cole R, Singh A, May P, Uc E, Dasgupta S, Narayanan N. Resting-state EEG measures cognitive impairment in Parkinson's disease. Res Sq [Preprint]. 2023 Mar 20:rs.3.rs-2666578. doi: 10.21203/rs.3.rs-2666578/v1. PMID 36993450
- [Background] Simmering JE, Welsh MJ, Schultz J, Narayanan NS. Use of Glycolysis-Enhancing Drugs and Risk of Parkinson's Disease. Mov Disord. 2022 Nov;37(11):2210-2216. doi: 10.1002/mds.29184. Epub 2022 Aug 22. PMID 36054705
- [Background] Cole RC, Okine DN, Yeager BE, Narayanan NS. Neuromodulation of cognition in Parkinson's disease. Prog Brain Res. 2022;269(1):435-455. doi: 10.1016/bs.pbr.2022.01.016. Epub 2022 Feb 11. PMID 35248205
- [Background] Cole RC, Espinoza AI, Singh A, Berger JI, Cavanagh JF, Wessel JR, Greenlee JD, Narayanan NS. Novelty-induced frontal-STN networks in Parkinson's disease. Cereb Cortex. 2022 Dec 20;33(2):469-485. doi: 10.1093/cercor/bhac078. PMID 35297483
- [Background] Espinoza AI, May P, Anjum MF, Singh A, Cole RC, Trapp N, Dasgupta S, Narayanan NS. A pilot study of machine learning of resting-state EEG and depression in Parkinson's disease. Clin Park Relat Disord. 2022 Sep 27;7:100166. doi: 10.1016/j.prdoa.2022.100166. eCollection 2022. PMID 36203748
- [Background] Zhang Q, Schultz JL, Aldridge GM, Simmering JE, Kim Y, Ogilvie AC, Narayanan NS. COVID-19 Case Fatality and Alzheimer's Disease. J Alzheimers Dis. 2021;84(4):1447-1452. doi: 10.3233/JAD-215161. PMID 34690147
- [Background] Singh A, Cole RC, Espinoza AI, Evans A, Cao S, Cavanagh JF, Narayanan NS. Timing variability and midfrontal ~4 Hz rhythms correlate with cognition in Parkinson's disease. NPJ Parkinsons Dis. 2021 Feb 15;7(1):14. doi: 10.1038/s41531-021-00158-x. PMID 33589640
- [Background] Groth CL, Singh A, Zhang Q, Berman BD, Narayanan NS. GABAergic Modulation in Movement Related Oscillatory Activity: A Review of the Effect Pharmacologically and with Aging. Tremor Other Hyperkinet Mov (N Y). 2021 Nov 10;11:48. doi: 10.5334/tohm.655. eCollection 2021. PMID 34824891
- [Background] Simmering JE, Welsh MJ, Liu L, Narayanan NS, Pottegard A. Association of Glycolysis-Enhancing alpha-1 Blockers With Risk of Developing Parkinson Disease. JAMA Neurol. 2021 Apr 1;78(4):407-413. doi: 10.1001/jamaneurol.2020.5157. PMID 33523098
- [Background] Zhang Q, Abdelmotilib H, Larson T, Keomanivong C, Conlon M, Aldridge GM, Narayanan NS. Cortical alpha-synuclein preformed fibrils do not affect interval timing in mice. Neurosci Lett. 2021 Nov 20;765:136273. doi: 10.1016/j.neulet.2021.136273. Epub 2021 Sep 30. PMID 34601038
- [Background] Anjum MF, Haug J, Alberico SL, Dasgupta S, Mudumbai R, Kennedy MA, Narayanan NS. Linear Predictive Approaches Separate Field Potentials in Animal Model of Parkinson's Disease. Front Neurosci. 2020 Apr 24;14:394. doi: 10.3389/fnins.2020.00394. eCollection 2020. PMID 32390797
- [Background] Singh A, Cole RC, Espinoza AI, Brown D, Cavanagh JF, Narayanan NS. Frontal theta and beta oscillations during lower-limb movement in Parkinson's disease. Clin Neurophysiol. 2020 Mar;131(3):694-702. doi: 10.1016/j.clinph.2019.12.399. Epub 2020 Jan 13. PMID 31991312
- [Background] Zhang Q, Schultz JL, Aldridge GM, Simmering JE, Narayanan NS. Coronavirus Disease 2019 Case Fatality and Parkinson's Disease. Mov Disord. 2020 Nov;35(11):1914-1915. doi: 10.1002/mds.28325. Epub 2020 Oct 15. No abstract available. PMID 32954522
- [Background] Zhang Q, Aldridge GM, Narayanan NS, Anderson SW, Uc EY. Approach to Cognitive Impairment in Parkinson's Disease. Neurotherapeutics. 2020 Oct;17(4):1495-1510. doi: 10.1007/s13311-020-00963-x. Epub 2020 Nov 17. PMID 33205381
- [Background] Anjum MF, Dasgupta S, Mudumbai R, Singh A, Cavanagh JF, Narayanan NS. Linear predictive coding distinguishes spectral EEG features of Parkinson's disease. Parkinsonism Relat Disord. 2020 Oct;79:79-85. doi: 10.1016/j.parkreldis.2020.08.001. Epub 2020 Aug 23. PMID 32891924
- [Background] Narayanan NS, Wessel JR, Greenlee JDW. The Fastest Way to Stop: Inhibitory Control and IFG-STN Hyperdirect Connectivity. Neuron. 2020 May 20;106(4):549-551. doi: 10.1016/j.neuron.2020.04.017. PMID 32437650
- [Background] Aldridge GM, Birnschein A, Denburg NL, Narayanan NS. Parkinson's Disease Dementia and Dementia with Lewy Bodies Have Similar Neuropsychological Profiles. Front Neurol. 2018 Mar 12;9:123. doi: 10.3389/fneur.2018.00123. eCollection 2018. PMID 29593630
- [Background] Singh A, Richardson SP, Narayanan N, Cavanagh JF. Mid-frontal theta activity is diminished during cognitive control in Parkinson's disease. Neuropsychologia. 2018 Aug;117:113-122. doi: 10.1016/j.neuropsychologia.2018.05.020. Epub 2018 May 23. PMID 29802866
- [Background] Kelley R, Flouty O, Emmons EB, Kim Y, Kingyon J, Wessel JR, Oya H, Greenlee JD, Narayanan NS. A human prefrontal-subthalamic circuit for cognitive control. Brain. 2018 Jan 1;141(1):205-216. doi: 10.1093/brain/awx300. PMID 29190362
- See also: Please send any questions about data to nandakumar-narayanan@uiowa.edu — https://narayanan.lab.uiowa.edu/home/data